CLINICAL TRIAL: NCT03215563
Title: Hybrid 18F-Fluoride Positron Emission Tomography-Magnetic Resonance Imaging in Patients With Acute Acute Neurovascular Syndrome
Brief Title: PET-MRI Imaging in Patients With Acute Neurovascular Syndrome
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: AC17058
Record Dates: First submitted 2017-06-14; First posted 2017-07-12 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Stroke; Carotid Stenosis
Keywords: atherosclerosis, imaging
MeSH Terms: conditions — Stroke; Carotid Stenosis; Atherosclerosis | interventions — Ultrasonography, Doppler, Transcranial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Carotid: Patients with carotid artery stenosis who either do not meet surgical criteria (< 50% by NASCET criteria for men, <70% for women), or meet criteria but do not undergo surgery (surgery declined or not offered) and are currently treated with OMT. This cohort will be recruited from the acute TIA clinics and Vascular Laboratory logbooks at Edinburgh Royal Infirmary and Western General Hospital.
  Interventions: Radiation: 18F PET-MRI; Diagnostic Test: Transcranial Doppler
- Non Carotid: Patients with an atherosclerotic disease in the aortic arch including origins of its major branches other than the internal carotid artery treated with OMT. Patients with a cardiac source of embolism will be excluded from the study. This group will be recruited from the acute TIA clinics and inpatients at Edinburgh Royal Infirmary and Western General Hospital.
  Interventions: Radiation: 18F PET-MRI; Diagnostic Test: Transcranial Doppler

INTERVENTIONS:
Radiation: 18F PET-MRI — 18F-fluoride Hybrid PET-MRI
Diagnostic Test: Transcranial Doppler — Microembolic Signals detection

SUMMARY:
Ischaemic stroke is a major cause of death and disability worldwide. In patients with recent stroke, the 18F-fluoride positron emission tomography-computed tomography highlights high-risk culprit carotid plaque and is more discriminatory than 18F-fluorodeoxyglucose. Using hybrid positron emission tomography-magnetic resonance imaging investigators propose to build upon these findings by prospectively assessing 18F-fluoride uptake in a broad range of patients with acute transient ischaemic attack or ischaemic stroke. Investigators will specifically examine the association of 18F-fluoride uptake with multiparametric magnetic resonance imaging assessments of atherosclerotic plaque, especially the role of thrombus and lipid. Finally, using transcranial Doppler and diffusion-weighted magnetic resonance brain imaging, an assessment of the functional consequences of 18F-fluoride-positive atherosclerotic plaque will be performed. If successful, this technique has a number of valuable translational applications including the better selection of patients for carotid intervention.

DETAILED DESCRIPTION:
The ability to identify the culprit carotid plaque represents a key goal in carotid artery imaging. Although an array of non-invasive imaging techniques can detect a wide spectrum of complementary high-risk characteristics, no single modality can reliably identify vulnerable plaques associated with future stroke development. Substantial histological data suggests that specific plaque components identify patients at high-risk for future ipsilateral stroke and cardiovascular events. This implies that investigators need to look beyond the traditional paradigm where the basis for carotid endarterectomy were formulated by an invasive imaging modality that provided no information on the arterial wall composition. Alternative imaging strategies are therefore required targeting not only in vivo carotid morphology but also plaque biology and disease activity. This is fundamental to optimal risk-stratification and appropriate selection of patients for high-risk vascular intervention. One new approach is to use non-invasive molecular imaging targeted at plaque biology using hybrid systems such as positron emission tomography-magnetic resonance imaging.

ELIGIBILITY:
Inclusion Criteria:

1. Patients above 40 years of age with carotid artery stenosis that do not achieve criteria for CEA (<50% for men, <70% for women, by NASCET criteria) or the patient has declined CEA.
2. Patients above 40 years of age with atherosclerotic disease of aortic arch and its branches.

Exclusion Criteria:

1. Patients with new stroke and a modified Rankin score >3
2. Chronic kidney disease with an estimated Glomerular Filtration Rate (eGFR) of <30 ml/min/1.73 m2
3. Atrial fibrillation
4. Pregnant women
5. Prior ipsilateral carotid intervention
6. Prior neck radiotherapy
7. Inability to tolerate the supine position
8. Participation in the study would result in delay to surgery
9. Psychiatric illness/social situations that would limit compliance with study requirements
10. History of allergic reaction attributed to 18F-Fluoride
11. History of allergic reaction to gadolinium contrast media
12. Metal implants or devices including pacemakers and defibrillators

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Two cohorts of patients with evidence of an acute stroke, transient ischaemic attack or amaurosis fugax will be recruited as early as possible, but within 14 days of symptom onset. All patients will undergo careful clinical evaluation including carotid Doppler ultrasound assessment and magnetic resonance imaging of the brain.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2017-10-12 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
18F-fluoride uptake in the culprit plaque in carotid, aortic and intra-cranial vessels. | 2 weeks
  18F-fluoride uptake will be measured by the mean and max Standardised Uptake Values (SUV) derived from the culprit atherosclerotic plaques.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Cardiovascular Science, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kaczynski J, Sellers S, Seidman MA, Syed M, Dennis M, Mcnaught G, Jansen M, Semple SI, Alcaide-Corral C, Tavares AAS, MacGillivray T, Debono S, Forsythe R, Tambyraja A, Slomka PJ, Leipsic J, Dweck MR, Whiteley W, Wardlaw J, van Beek EJR, Newby DE, Williams MC. 18F-NaF PET/MRI for Detection of Carotid Atheroma in Acute Neurovascular Syndrome. Radiology. 2022 Oct;305(1):137-148. doi: 10.1148/radiol.212283. Epub 2022 Jun 7. PMID 35670715